CLINICAL TRIAL: NCT06432127
Title: Role of Ultrasound Guide Greater Occipital Nerve Block at Second Cervical Vertebra in Migraine Headache Prophylaxis in Patients With Failed Oral Prophylaxis Medication : A Randomized Controlled Study in Thailand
Brief Title: Role of Ultrasound Guide Greater Occipital Nerve Block at Second Cervical Vertebra in Migraine Headache Prophylaxis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 256/2024
Record Dates: First submitted 2024-05-15; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Use Normal saline 3 ml as the injection agent
  Interventions: Drug: Placebo
- Bupivacaine (Experimental): Use 0.5% Bupivacaine 3ml as the injection agent
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Placebo — Unilateral Greater occipital nerve block at C2 level under ultrasound guide with needle in plane technique during ultrasound using normal saline 3 mL
  Arms: Placebo
Drug: Bupivacaine — Unilateral Greater occipital nerve block at C2 level under ultrasound guide with needle in plane technique during ultrasound using 0.5% Bupivacaine 3 mL
  Arms: Bupivacaine

SUMMARY:
The goal of this randomized controlled study in Thailand. is to find if there is a role of local anesthetic greater occipital nerve block at Cervical spine level 2 under ultrasound guide in prophylaxis of episodic migraine and chronic migraine in patients with failed oral prophylaxis medication.

According to guidelines of the International Headache Society for controlled trials of preventive treatment of migraine attacks in episodic and chronic migraine,the primary and secondary outcome were monitoring followed by these research guideline

After informed consent, volunteer will be stratified random into 2 groups of injection agent at unilateral greater occipital nerve block on headache site under US guide by pain physician

* Normal saline
* 0.5% bupivacaine the injection was done 2 times between Week 0 and week 4 as to wean off placebo effect the volunteer will be monitor by pain diary at 1 month before intervention at week 0,4,8,12 and follow up at week 24 for Migraine Disability Assessment Test (MIDAS) ,Thai Hospital-Anxiety-depression index(Thai-HADS)

DETAILED DESCRIPTION:
* Neurologist screening candidate volunteers for this study, following the inclusion and exclusion criteria
* Candidate volunteers attended pain clinic for he protocol detail about this research and informed consent
* After signing consent, Volunteers would be stratified randomization into 2 groups between Normal saline and bupivacaine
* Volunteers would be done base line headache diary for 1 month before performing the procedure (Week -4 to week0)
* At Week 0, Volunteers would be applied local anesthetic cream at skin injection site before done the procedure
* According to stratified randomization, Pain interventionist and also volunteers would be blinded to the group
* First Unilateral greater occipital nerve block at Cervical spine level 2 (C2) was done under ultrasound guide (Week0)
* Telemedicine Follow up at week 2
* Second Unilateral greater occipital nerve block at C2 level was done under ultrasound guide (Week4)
* Volunteers would be follow up via telemedicine and done headache diary until 3 months after 1st injection
* Volunteers would be follow up according to outcome monitoring protocol in Week 0,4,8,12,24

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 -65 years old
2. Diagnosis as episodic migraine or chronic migraine and had indication to use migraine prophylaxis
3. Volunteer prefer to use research procedure as first choice of migraine prophylaxis
4. Volunteer already had migraine prophylaxis treatment but still has the one of these following problem 4.1 Frequency of migraine attack more than 4 times/month 4.2 Severe migraine headache & disturb daily life in spite of using migraine prophylaxis 4.3 Having migraine medication side effect, either from prophylaxis or acute attack medication and cannot titration medication dosage 4.4 migraine attack not improved as using many migraine prophylaxis medications 4.5 Having contra-indication to use prophylaxis migraine medication or standard prophylaxis procedure such as botulinum toxin 4.6 Cannot take prophylaxis medication daily (low compliance) 4.7 Had financial problems in using standard prophylaxis migraine medication or procedure 4.8 Medication overuse headache

Exclusion Criteria:

1. Had these type of headache in combination with migraine

   * cervicogenic headache
   * occipital neuralgia
   * secondary headache
2. Had contraindication on greater occipital nerve block injection at cervical spine level 2 under ultrasound-guided such as skin infection in needle site
3. Allergy to local anesthetic
4. Uncontrolled psychiatric disorder in 3 months before attending research
5. Cannot understand or reading, writing Thai language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
change of Frequency headache day /month | at Week 0,4,8,12,24 compared to base line at 1 months before injection procedure
  by using headache diary
change of migraine attack day /month from headache diary | at Week 0,4,8,12,24 compared to base line at 1 months before injection procedure
  by using headache diary

SECONDARY OUTCOMES:
change in severity of headache day per month (decrease of moderate-severe pain) | at Week 0,4,8,12,24 compared to base line at 1 months before injection procedure
  decrease of moderate-severe pain day per month compare to baseline by using headache diary
Thai-Migraine Disability Assessment | at Week 12,24 compare to baseline
  Thai-Migraine Disability Assessment (MIDAS) ,Score 0 to 21+ ( 0-5 marks = little or no disability and more than 21+ =severe disability
Thai-Hospital Anxiety and Depression Scale | at Week 0,4,8,12,24 compared to base line at 1 months before injection procedure
  Thai-Hospital Anxiety and Depression Scale (Thai HADS) , divided into anxiety and depression part ,if either of the score in each depression or anxiety more than 11 mean abnormal
Healthcare outcomes/quality of life | at Week 0,4,8,12,24 compared to base line at 1 months before injection procedure
  by EuroQoL- (EQ-5D) measured health-related quality of life with 5 dimension (mobility, health care, usual activity, Pain, Anxiety/depression and in each of them had 5 grading 1-5 by 1 means no problem and 5 means extreme problem) after having score in each dimension, calculated utility score would be done
Patient's reported outcome measurement (PGI-C) | at Week 0,4,8,12,24 compared to base line at 1 months before injection procedure
  Patient's reported outcome measurement (PGI-C), score grading 1-7 by 1 very much worse to very much improved , 7 means very much worse

CONTACTS AND LOCATIONS:
Overall Officials: RAVIWON ATISOOK, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Raviwon Atisook, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
will be consider again after data collection